CLINICAL TRIAL: NCT00077974
Title: A Pivotal Study Of SU011248 In The Treatment Of Patients With Cytokine-Refractory Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181006; NCT00082849 (obsolete NCT alias)
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Results first posted 2009-11-03 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: SU011248 — 50-mg orally taken daily for 4 weeks and off treatment for 2 weeks until progression or unacceptable toxicity
  Other Names: Sunitinib, SUTENT

SUMMARY:
To assess the safety and efficacy of SU011248 in patients with metastatic, refractory renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Cytokine refractory metastatic renal cell carcinoma with clear cell component
* Radiographic evidence of disease progression during or within 9 months of completion of 1 cytokine therapy
* Prior nephrectomy

Exclusion Criteria:

* Prior treatment with any systemic therapy other than 1 cytokine therapy
* History of or known brain metastases
* Uncontrolled hypertension or other significant cardiac events within the 12 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2004-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Motzer RJ, Rini BI, Bukowski RM, Curti BD, George DJ, Hudes GR, Redman BG, Margolin KA, Merchan JR, Wilding G, Ginsberg MS, Bacik J, Kim ST, Baum CM, Michaelson MD. Sunitinib in patients with metastatic renal cell carcinoma. JAMA. 2006 Jun 7;295(21):2516-24. doi: 10.1001/jama.295.21.2516. PMID 16757724
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181006&StudyName=A%20Pivotal%20Study%20Of%20SU011248%20In%20The%20Treatment%20Of%20Patients%20With%20Cytokine-Refractory%20Metastatic%20Renal%20Cell%20Carcinoma.%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Malate: 50 milligrams per day on Schedule 4/2 (4 weeks daily treatment followed by 2 weeks off treatment in repeated 6-week cycles)
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 106
Completed | 2
Not Completed | 104
Not completed — Adverse Event | 22
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 76
Not completed — Decision of Sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
Age, Customized [Number; unit: participants]
  < 65 years | 87
  >= 65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)
Description: Overall confirmed objective response = confirmed Complete Response (CR) or confirmed Partial Response (PR) according to RECIST. CR defined as disappearance of all target lesions. PR defined as >= 30 percent decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From start of study treatment until Day 28 of Cycles 1-5, Day 28 of even Cycles thereafter
Population: The intent-to-treat (ITT) population included all subjects who enrolled in the study that received at least 1 dose of study medication. This was the primary population for all efficacy analyses and safety analyses.
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
participants | 35
Statistical Analysis 1: Comparison: Sunitinib Malate; Test type: Superiority or Other; Percent = 33, 95% CI [24.2 to 42.8] — Using exact method based on binomial distribution. Percent equals n divided by N times 100

2. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]).
Time Frame: From start of study treatment until Day 28 of Cycles 1-5, Day 28 of even Cycles thereafter
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
weeks | 46.3 [34.0 to 58.9]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7.
  DR was calculated for the subgroup of patients with a confirmed objective tumor response.
Time Frame: Day 28 of Cycles 1-5, Day 28 of even Cycles thereafter or death due to cancer
Population: ITT subgroup of patients with a confirmed objective tumor response
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 35
weeks | 60.4 [48.4 to 70.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the subject current status was death).
Time Frame: From start of study treatment until death
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
weeks | 104.1 [61.0 to 133.1]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: From start of study treatment until Day 28 of Cycles 1-5, Day 28 of even Cycles thereafter or death
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
weeks | 38.0 [33.9 to 58.4]

6. Secondary Outcome: Percent Chance of Patient Survival
Description: Probability of survival 1 year and 2 years after the first dose of study treatment
Time Frame: From start of study treatment until death
Population: ITT
Measure: Number; unit: percent chance of survival
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
percent chance of survival
  1 year | 67.2
  2 years | 50.2

7. Secondary Outcome: Observed Plasma Trough Concentrations of Sunitinib
Description: Observed plasma trough (predose) (Cmin) concentrations of sunitinib
Time Frame: Day 28 of Cycle 1 through 4, Day 1 of Cycles 5 and greater
Population: Pharmacokinetic analysis population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 104
nanograms per milliliter
  Cycle 1 Day 28 (n = 103) | 46.82 (24.19)
  Cycle 2 Day 28 (n = 81) | 50.13 (24.66)
  Cycle 3 Day 28 (n = 73) | 49.36 (25.26)
  Cycle 4 Day 28 (n = 66) | 53.18 (22.62)
  Cycle 5 Day 1 (n = 63) | 1.55 (1.48)
  Cycle 6 Day 1 (n = 59) | 1.44 (1.37)
  Cycle 7 Day 1 (n = 52) | 1.51 (1.90)
  Cycle 8 Day 1 (n = 48) | 1.60 (1.38)
  Cycle 9 Day 1 (n = 46) | 1.60 (1.58)
  Cycle 10 Day 1 (n = 41) | 1.69 (1.97)
  Cycle 11 Day 1 (n = 38) | 2.05 (3.00)
  Cycle 12 Day 1 (n = 34) | 1.72 (1.66)
  Cycle 13 Day 1 (n = 30) | 1.74 (1.57)
  Cycle 14 Day 1 (n = 30) | 1.60 (1.45)
  Cycle 15 Day 1 (n = 24) | 1.56 (2.17)
  Cycle 16 Day 1 (n = 24) | 1.46 (1.23)
  Cycle 17 Day 1 (n = 19) | 1.42 (1.65)
  Cycle 18 Day 1 (n = 16) | 2.20 (2.17)
  Cycle 19 Day 1 (n = 14) | 1.34 (1.18)
  Cycle 20 Day 1 (n = 12) | 2.96 (3.53)
  Cycle 21 Day 1 (n = 11) | 2.53 (2.07)
  Cycle 22 Day 1 (n = 11) | 2.18 (2.57)
  Cycle 23 Day 1 (n = 7) | 3.14 (2.70)
  Cycle 24 Day 1 (n = 7) | 2.75 (1.86)
  Cycle 25 Day 1 (n = 6) | 1.99 (1.37)
  Cycle 26 Day 1 (n = 6) | 2.46 (2.43)
  Cycle 27 Day 1 (n = 6) | 1.20 (1.21)
  Cycle 28 Day 1 (n = 4) | 1.75 (1.61)
  Cycle 29 Day 1 (n = 5) | 2.93 (3.64)
  Cycle 30 Day 1 (n = 4) | 1.02 (0.90)

8. Secondary Outcome: Observed Plasma Trough Concentrations of Sunitinib Metabolite
Description: Observed plasma trough (predose) (Cmin) concentrations of sunitinib metabolite (SU012662)
Time Frame: Day 28 of Cycle 1 through 4, Day 1 of Cycles 5 and greater
Population: Pharmacokinetic analysis population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
nanograms per milliliter
  Cycle 1 Day 28 (n = 103) | 26.44 (15.66)
  Cycle 2 Day 28 (n = 81) | 28.21 (17.21)
  Cycle 3 Day 28 (n = 73) | 28.32 (18.38)
  Cycle 4 Day 28 (n = 66) | 28.54 (16.93)
  Cycle 5 Day 1 (n = 63) | 2.50 (1.60)
  Cycle 6 Day 1 (n = 59) | 2.64 (1.67)
  Cycle 7 Day 1 (n = 52) | 2.64 (1.98)
  Cycle 8 Day 1 (n = 48) | 2.66 (1.68)
  Cycle 9 Day 1 (n = 46) | 2.81 (2.32)
  Cycle 10 Day 1 (n = 41) | 2.54 (1.87)
  Cycle 11 Day 1 (n = 38) | 2.78 (3.40)
  Cycle 12 Day 1 (n = 34) | 2.67 (2.29)
  Cycle 13 Day 1 (n = 30) | 2.77 (2.03)
  Cycle 14 Day 1 (n = 30) | 2.49 (2.05)
  Cycle 15 Day 1 (n = 24) | 2.51 (2.98)
  Cycle 16 Day 1 (n = 24) | 2.30 (1.84)
  Cycle 17 Day 1 (n = 19) | 1.83 (1.49)
  Cycle 18 Day 1 (n = 16) | 2.16 (1.07)
  Cycle 19 Day 1 (n = 14) | 2.06 (1.82)
  Cycle 20 Day 1 (n = 12) | 2.92 (1.86)
  Cycle 21 Day 1 (n = 11) | 3.13 (2.19)
  Cycle 22 Day 1 (n = 11) | 3.24 (3.12)
  Cycle 23 Day 1 (n = 7) | 3.10 (2.25)
  Cycle 24 Day 1 (n = 7) | 2.64 (1.68)
  Cycle 25 Day 1 (n = 6) | 1.99 (1.07)
  Cycle 26 Day 1 (n = 6) | 2.60 (2.26)
  Cycle 27 Day 1 (n = 6) | 1.36 (1.22)
  Cycle 28 Day 1 (n = 4) | 1.81 (1.20)
  Cycle 29 Day 1 (n = 5) | 2.43 (2.12)
  Cycle 30 Day 1 (n = 4) | 1.10 (0.73)

9. Secondary Outcome: Observed Plasma Trough Concentrations of Sunitinib Plus Metabolite
Description: Observed plasma trough (predose) concentrations of sunitinib plus its metabolite (SU012662)
Time Frame: Day 28 of Cycle 1 through 4, Day 1 of Cycles 5 and greater
Population: Pharmacokinetic analysis population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
nanograms per milliliter
  Cycle 1 Day 28 (n = 103) | 73.26 (36.85)
  Cycle 2 Day 28 (n = 81) | 78.34 (39.03)
  Cycle 3 Day 28 (n = 73) | 77.68 (39.84)
  Cycle 4 Day 28 (n = 66) | 81.71 (36.55)
  Cycle 5 Day 1 (n = 63) | 4.04 (2.80)
  Cycle 6 Day 1 (n = 59) | 4.08 (2.72)
  Cycle 7 Day 1 (n = 52) | 4.15 (3.57)
  Cycle 8 Day 1 (n = 48) | 4.26 (2.78)
  Cycle 9 Day 1 (n = 46) | 4.41 (3.65)
  Cycle 10 Day 1 (n = 41) | 4.23 (3.69)
  Cycle 11 Day 1 (n = 38) | 4.83 (6.34)
  Cycle 12 Day 1 (n = 34) | 4.39 (3.69)
  Cycle 13 Day 1 (n = 30) | 4.52 (3.36)
  Cycle 14 Day 1 (n = 30) | 4.09 (3.37)
  Cycle 15 Day 1 (n = 24) | 4.07 (5.00)
  Cycle 16 Day 1 (n = 24) | 3.75 (2.63)
  Cycle 17 Day 1 (n = 19) | 3.25 (3.03)
  Cycle 18 Day 1 (n = 16) | 4.35 (2.90)
  Cycle 19 Day 1 (n = 14) | 3.40 (2.87)
  Cycle 20 Day 1 (n = 12) | 5.88 (5.19)
  Cycle 21 Day 1 (n = 11) | 5.66 (4.09)
  Cycle 22 Day 1 (n = 11) | 5.43 (5.61)
  Cycle 23 Day 1 (n = 7) | 6.24 (4.78)
  Cycle 24 Day 1 (n = 7) | 5.39 (3.31)
  Cycle 25 Day 1 (n = 6) | 3.97 (2.32)
  Cycle 26 Day 1 (n = 6) | 5.06 (4.61)
  Cycle 27 Day 1 (n = 6) | 2.55 (2.41)
  Cycle 28 Day 1 (n = 4) | 3.56 (2.77)
  Cycle 29 Day 1 (n = 5) | 5.36 (5.74)
  Cycle 30 Day 1 (n = 4) | 2.13 (1.57)

10. Secondary Outcome: Dose Corrected Plasma Trough Concentrations of Sunitinib
Description: Dose corrected plasma trough (predose) (Cmin) concentrations of sunitinib. Dose-corrected trough concentrations were set to missing for trough samples collected outside acceptable times from dose administration, samples not collected within scheduled day range, samples with missing collection or administration dates or times, samples collected with dose interruption, and samples collected with inconsistent dose level within 10 days of last dose date.
Time Frame: Day 28 of Cycle 1 through 4, Day 1 of Cycles 5 and greater
Population: Pharmacokinetic analysis population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
nanograms per milliliter
  Cycle 1 Day 28 (n = 33) | 53.64 (22.54)
  Cycle 2 Day 28 (n = 26) | 55.94 (25.52)
  Cycle 3 Day 28 (n = 20) | 69.44 (33.21)
  Cycle 4 Day 28 (n = 25) | 64.33 (41.46)
  Cycle 5 Day 1 (n = 28) | 1.94 (3.24)
  Cycle 6 Day 1 (n = 41) | 2.15 (2.94)
  Cycle 7 Day 1 (n = 35) | 2.04 (4.10)
  Cycle 8 Day 1 (n = 32) | 2.32 (2.77)
  Cycle 9 Day 1 (n = 32) | 2.07 (2.62)
  Cycle 10 Day 1 (n = 32) | 2.68 (4.32)
  Cycle 11 Day 1 (n = 25) | 3.42 (6.86)
  Cycle 12 Day 1 (n = 28) | 1.94 (1.63)
  Cycle 13 Day 1 (n = 23) | 2.23 (2.49)
  Cycle 14 Day 1 (n = 24) | 2.41 (2.46)
  Cycle 15 Day 1 (n = 16) | 1.58 (1.09)
  Cycle 16 Day 1 (n = 18) | 2.42 (2.48)
  Cycle 17 Day 1 (n = 17) | 2.23 (2.66)
  Cycle 18 Day 1 (n = 14) | 3.05 (4.57)
  Cycle 19 Day 1 (n = 11) | 1.92 (1.58)
  Cycle 20 Day 1 (n = 11) | 5.09 (7.47)
  Cycle 21 Day 1 (n = 8) | 3.41 (3.24)
  Cycle 22 Day 1 (n = 9) | 3.91 (5.45)
  Cycle 23 Day 1 (n = 6) | 4.53 (3.89)
  Cycle 24 Day 1 (n = 6) | 3.82 (3.68)
  Cycle 25 Day 1 (n = 5) | 3.14 (3.24)
  Cycle 26 Day 1 (n = 5) | 4.09 (5.70)
  Cycle 27 Day 1 (n = 5) | 2.12 (2.58)
  Cycle 28 Day 1 (n = 4) | 2.97 (3.36)
  Cycle 29 Day 1 (n = 4) | 4.02 (5.60)
  Cycle 30 Day 1 (n = 3) | 1.36 (1.50)

11. Secondary Outcome: Dose Corrected Plasma Trough Concentrations of Sunitinib Metabolite
Description: Dose corrected plasma trough (predose) (Cmin) concentrations of sunitinib metabolite (SU012662). Dose-corrected trough concentrations were set to missing for trough samples collected outside acceptable times from dose administration, samples not collected within scheduled day range, samples with missing collection or administration dates or times, samples collected with dose interruption, and samples collected with inconsistent dose level within 10 days of last dose date.
Time Frame: Day 28 of Cycle 1 through 4, Day 1 of Cycles 5 and greater
Population: Pharmacokinetic analysis population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
nanograms per milliliter
  Cycle 1 Day 28 (n = 33) | 31.85 (18.15)
  Cycle 2 Day 28 (n = 26) | 28.15 (19.80)
  Cycle 3 Day 28 (n = 20) | 40.53 (20.38)
  Cycle 4 Day 28 (n = 25) | 38.04 (24.29)
  Cycle 5 Day 1 (n = 28) | 2.99 (2.55)
  Cycle 6 Day 1 (n = 41) | 3.35 (2.52)
  Cycle 7 Day 1 (n = 35) | 3.11 (3.13)
  Cycle 8 Day 1 (n = 32) | 3.37 (2.34)
  Cycle 9 Day 1 (n = 32) | 3.45 (2.80)
  Cycle 10 Day 1 (n = 32) | 3.61 (3.62)
  Cycle 11 Day 1 (n = 25) | 4.37 (8.13)
  Cycle 12 Day 1 (n = 28) | 3.24 (2.82)
  Cycle 13 Day 1 (n = 23) | 3.68 (2.79)
  Cycle 14 Day 1 (n = 24) | 3.54 (2.60)
  Cycle 15 Day 1 (n = 16) | 2.80 (1.82)
  Cycle 16 Day 1 (n = 18) | 3.40 (2.27)
  Cycle 17 Day 1 (n = 17) | 2.55 (2.23)
  Cycle 18 Day 1 (n = 14) | 2.59 (1.69)
  Cycle 19 Day 1 (n = 11) | 2.93 (2.33)
  Cycle 20 Day 1 (n = 11) | 4.53 (3.82)
  Cycle 21 Day 1 (n = 8) | 3.97 (2.78)
  Cycle 22 Day 1 (n = 9) | 5.31 (6.73)
  Cycle 23 Day 1 (n = 6) | 4.26 (3.16)
  Cycle 24 Day 1 (n = 6) | 3.62 (2.49)
  Cycle 25 Day 1 (n = 5) | 3.00 (2.18)
  Cycle 26 Day 1 (n = 5) | 4.49 (5.29)
  Cycle 27 Day 1 (n = 5) | 2.36 (2.57)
  Cycle 28 Day 1 (n = 4) | 2.94 (2.63)
  Cycle 29 Day 1 (n = 4) | 3.32 (3.28)
  Cycle 30 Day 1 (n = 3) | 1.18 (1.08)

12. Secondary Outcome: Dose Corrected Plasma Trough Concentrations of Sunitinib Plus Metabolite
Description: Dose corrected plasma trough (predose) (Cmin) concentrations of sunitinib plus its metabolite (SU012662). Dose-corrected trough concentrations were set to missing for trough samples collected outside acceptable times from dose administration, samples not collected within scheduled day range, samples with missing collection or administration dates or times, samples collected with dose interruption, and samples collected with inconsistent dose level within 10 days of last dose date.
Time Frame: Day 28 of Cycle 1 through 4, Day 1 of Cycles 5 and greater
Population: Pharmacokinetic analysis population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 106
nanograms per milliliter
  Cycle 1 Day 28 (n = 33) | 85.49 (37.49)
  Cycle 2 Day 28 (n = 26) | 84.09 (42.11)
  Cycle 3 Day 28 (n = 20) | 109.97 (48.38)
  Cycle 4 Day 28 (n = 25) | 102.37 (62.69)
  Cycle 5 Day 1 (n = 28) | 4.93 (5.49)
  Cycle 6 Day 1 (n = 41) | 5.50 (5.14)
  Cycle 7 Day 1 (n = 35) | 5.15 (6.97)
  Cycle 8 Day 1 (n = 32) | 5.69 (4.86)
  Cycle 9 Day 1 (n = 32) | 5.52 (5.22)
  Cycle 10 Day 1 (n = 32) | 6.29 (7.80)
  Cycle 11 Day 1 (n = 25) | 7.78 (14.94)
  Cycle 12 Day 1 (n = 28) | 5.19 (4.08)
  Cycle 13 Day 1 (n = 23) | 5.91 (5.03)
  Cycle 14 Day 1 (n = 24) | 5.95 (4.80)
  Cycle 15 Day 1 (n = 16) | 4.39 (2.48)
  Cycle 16 Day 1 (n = 18) | 5.82 (4.21)
  Cycle 17 Day 1 (n = 17) | 4.78 (4.79)
  Cycle 18 Day 1 (n = 14) | 5.64 (6.01)
  Cycle 19 Day 1 (n = 11) | 4.85 (3.77)
  Cycle 20 Day 1 (n = 11) | 9.63 (11.00)
  Cycle 21 Day 1 (n = 8) | 7.38 (5.80)
  Cycle 22 Day 1 (n = 9) | 9.23 (12.13)
  Cycle 23 Day 1 (n = 6) | 8.79 (6.77)
  Cycle 24 Day 1 (n = 6) | 7.44 (5.84)
  Cycle 25 Day 1 (n = 5) | 6.13 (5.29)
  Cycle 26 Day 1 (n = 5) | 8.58 (10.94)
  Cycle 27 Day 1 (n = 5) | 4.48 (5.14)
  Cycle 28 Day 1 (n = 4) | 5.90 (5.96)
  Cycle 29 Day 1 (n = 4) | 7.34 (8.85)
  Cycle 30 Day 1 (n = 3) | 2.54 (2.58)

ADVERSE EVENTS:
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 46/106
Other Adverse Events (participants affected / at risk) | 106/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=106)
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Disease progression (General disorders) | 7
Fatigue (General disorders) | 1
Impaired healing (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Abscess (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Pancreatic abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Ejection fraction decreased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Convulsion (Nervous system disorders) | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 2
Ureteric obstruction (Renal and urinary disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Fracture treatment (Surgical and medical procedures) | 1
Tumour excision (Surgical and medical procedures) | 1
Aortic stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=106)
Anaemia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Hypothyroidism (Endocrine disorders) | 21
Lacrimation increased (Eye disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 19
Abdominal pain upper (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 40
Diarrhoea (Gastrointestinal disorders) | 67
Dry mouth (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 49
Dysphagia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12
Glossodynia (Gastrointestinal disorders) | 11
Haematochezia (Gastrointestinal disorders) | 6
Haemorrhoids (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 66
Oral pain (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 43
Vomiting (Gastrointestinal disorders) | 51
Chest discomfort (General disorders) | 7
Chest pain (General disorders) | 18
Chills (General disorders) | 20
Fatigue (General disorders) | 84
Mucosal inflammation (General disorders) | 28
Oedema (General disorders) | 10
Oedema peripheral (General disorders) | 22
Pain (General disorders) | 13
Pyrexia (General disorders) | 19
Nasopharyngitis (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 22
Urinary tract infection (Infections and infestations) | 9
Aspartate aminotransferase increased (Investigations) | 6
Blood creatinine increased (Investigations) | 9
Ejection fraction decreased (Investigations) | 19
Haemoglobin decreased (Investigations) | 8
Lipase increased (Investigations) | 12
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 16
Weight decreased (Investigations) | 18
Weight increased (Investigations) | 7
White blood cell count decreased (Investigations) | 12
Anorexia (Metabolism and nutrition disorders) | 43
Dehydration (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 13
Flank pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37
Dizziness (Nervous system disorders) | 19
Dysgeusia (Nervous system disorders) | 54
Headache (Nervous system disorders) | 32
Hypoaesthesia (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 10
Peripheral sensory neuropathy (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 14
Dysuria (Renal and urinary disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 14
Blister (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 23
Erythema (Skin and subcutaneous tissue disorders) | 15
Hair colour changes (Skin and subcutaneous tissue disorders) | 21
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 30
Periorbital oedema (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 38
Skin discolouration (Skin and subcutaneous tissue disorders) | 35
Skin exfoliation (Skin and subcutaneous tissue disorders) | 12
Skin lesion (Skin and subcutaneous tissue disorders) | 10
Skin reaction (Skin and subcutaneous tissue disorders) | 8
Hot flush (Vascular disorders) | 7
Hypertension (Vascular disorders) | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.